CLINICAL TRIAL: NCT07066319
Title: Impact of Gait Training on Lower Extremity Motor Function and Balance Performance in Stroke Survivors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Hamna Sarfraz, Research Associate, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-UOL-SMC/001-36/2024
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke Rehabilitation; Gait Training; Proprioceptive Neuromuscular Facilitation (PNF); Conventional Physical Therapy; Motor Recovery; Balance Training; Functional Independence; Fugl-Meyer Assessment; Berg Balance Scale; Wisconsin Gait Scale; Functional Independence Measure (FIM); Lower Limb Motor Function; Neurorehabilitation; Stroke Survivors; Physiotherapy
MeSH Terms: conditions — Stroke | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel intervention groups. Each group will receive a different physiotherapy protocol without crossover between arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gait Training with Proprioceptive Neuromuscular Facilitation (PNF) (Experimental): Participants in this arm will receive gait training integrated with Proprioceptive Neuromuscular Facilitation (PNF) techniques. The intervention will be delivered over 12 weeks, with sessions lasting 45 minutes, three times per week. Each session includes a 10-minute warm-up, 30 minutes of PNF-based gait training involving diagonal movement patterns and resistance exercises, and a 5-minute cool-down. Manual resistance and verbal cueing will be used to promote motor control, postural alignment, and dynamic stability.
  Interventions: Behavioral: Gait Training with Proprioceptive Neuromuscular Facilitation (PNF)
- Gait Training with Conventional Physical Therapy (Experimental): Participants in this group will receive structured gait training alongside conventional physiotherapy techniques. Sessions will be conducted three times per week for 12 weeks, each lasting 45 minutes. The protocol includes a 10-minute warm-up with flexibility and balance activities, 30 minutes of gait-focused exercises (e.g., step training, overground walking), and a 5-minute cool-down. Conventional PT methods such as strengthening, ROM exercises, and functional mobility drills will be used to improve gait performance and lower limb function.
  Interventions: Behavioral: Gait Training with Conventional Physiotherapy
- Combined PNF and Conventional Physiotherapy (Experimental): This group will receive a hybrid intervention combining Proprioceptive Neuromuscular Facilitation (PNF) and conventional physiotherapy techniques. Each session will last 45 minutes, three times per week for 12 weeks. The intervention includes a 10-minute PNF warm-up, 25 minutes of integrated gait training and functional exercises (balance, strengthening, mobility), and a 10-minute cool-down. The goal is to maximize motor recovery, neuromuscular coordination, and balance in stroke survivors.
  Interventions: Behavioral: Combined PNF and Conventional Physiotherapy (without direct gait training)

INTERVENTIONS:
Behavioral: Gait Training with Proprioceptive Neuromuscular Facilitation (PNF) — A physiotherapeutic intervention combining structured gait training with Proprioceptive Neuromuscular Facilitation (PNF) techniques. Sessions include rhythmic initiation, diagonal movement patterns, and resistance-based facilitation to enhance lower limb motor control and balance in stroke survivors. Delivered 3 times/week for 12 weeks, 45 minutes per session.
  Other Names: PNF Gait Therapy; Neuromuscular Gait Facilitation
  Arms: Gait Training with Proprioceptive Neuromuscular Facilitation (PNF)
Behavioral: Gait Training with Conventional Physiotherapy — A rehabilitation protocol integrating traditional gait training (step drills, overground walking) with conventional physiotherapy exercises focused on lower limb strength, range of motion, and postural balance. Conducted over 12 weeks, 3 sessions per week, 45 minutes each.
  Other Names: CPT Gait Training; Standard Physiotherapy for Stroke
  Arms: Gait Training with Conventional Physical Therapy
Behavioral: Combined PNF and Conventional Physiotherapy (without direct gait training) — This intervention blends Proprioceptive Neuromuscular Facilitation (PNF) with conventional physiotherapy, excluding dedicated gait tasks. It includes rhythmic stabilization, functional mobility drills, and resistance-based exercises aimed at improving neuromuscular re-education, balance, and independence. Delivered 3 times/week for 12 weeks, 45 minutes per session.
  Other Names: PNF+CPT Stroke Rehab; Hybrid Motor Recovery Therapy
  Arms: Combined PNF and Conventional Physiotherapy

SUMMARY:
This randomized clinical trial evaluates and compares the effectiveness of three physiotherapy-based rehabilitation strategies in improving gait, motor function, balance, and independence in individuals recovering from stroke. Stroke survivors often face challenges such as impaired walking, weak lower limbs, and poor postural control. Combining targeted interventions such as Proprioceptive Neuromuscular Facilitation (PNF) and Conventional Physical Therapy (CPT) may enhance functional outcomes.

Ninety-nine participants were randomly assigned to one of three groups:

Group A received Gait Training with PNF.

Group B received Gait Training with Conventional Physiotherapy.

Group C received a hybrid intervention combining PNF and Conventional Physiotherapy.

All interventions were delivered over 12 weeks, in 45-minute sessions conducted three times per week. Assessments were conducted at baseline, 3 weeks, and 6 weeks post-intervention.

The study used validated tools to measure progress in walking quality (Wisconsin Gait Scale - WGS), lower limb motor recovery (Fugl-Meyer Assessment - FMA-LE), balance (Berg Balance Scale - BBS), and daily functional ability (Functional Independence Measure - FIM).

To enable in-depth analysis, six outcome domains were created by combining different pairs of these tools:

A1: WGS + FMA-LE + FIM + BBS (overall recovery)

A2: WGS + BBS (gait and balance)

A3: WGS + FMA-LE (gait and motor recovery)

A4: BBS + FMA-LE (balance and motor recovery)

A5: WGS + FIM (gait and functional independence)

A6: BBS + FIM (balance and independence)

This study aims to identify the most effective rehabilitation strategy among the three to support physical recovery and improve independence in post-stroke individuals.

DETAILED DESCRIPTION:
This randomized clinical trial was conducted to investigate the comparative effects of three distinct gait-focused rehabilitation protocols on lower extremity motor function, balance performance, and functional independence in stroke survivors. The trial was carried out at the Department of Physiotherapy, Sehat Medical Complex, Hanjarwal, Lahore, over six months, following ethical approval.

A total sample of 99 participants was determined using G*Power, accounting for a 15% dropout rate. The participants were randomly allocated to one of three intervention groups (n=33 per group). Inclusion criteria required participants to be aged 40-80 years, have a confirmed diagnosis of stroke (ischemic or hemorrhagic), be at least 3 months post-stroke, and capable of understanding commands (GCS ≥ 9). Exclusion criteria included history of multiple strokes, significant comorbidities, or severe mobility or cognitive limitations.

Intervention Groups:

Group A (Gait Training + PNF):

45-minute sessions, 3 times per week for 12 weeks, combining dynamic gait training with PNF techniques such as diagonal movement patterns, rhythmic initiation, and manual resistance to enhance neuromuscular control and coordination.

Group B (Gait Training + Conventional Physiotherapy):

Participants underwent overground walking, step drills, strength and balance exercises, sit-to-stand transitions, and joint mobilizations to improve postural control, muscle strength, and walking pattern.

Group C (PNF + Conventional Physiotherapy):

This group received PNF-based resistance and rhythmic stabilization along with traditional exercises (e.g., mobility drills, resistance training, flexibility work), excluding direct gait training.

Each protocol targeted specific recovery domains, progressing in intensity and complexity over time. Functional and motor outcomes were assessed using:

Wisconsin Gait Scale (WGS) for gait performance

Fugl-Meyer Assessment - Lower Extremity (FMA-LE) for motor recovery

Berg Balance Scale (BBS) for balance assessment

Functional Independence Measure (FIM) for daily functional capability

To allow for a comprehensive evaluation, outcome data were analyzed under six analytical combinations:

A1: All four measures combined (WGS, FMA-LE, FIM, BBS)

A2: Gait and balance (WGS + BBS)

A3: Gait and motor recovery (WGS + FMA-LE)

A4: Balance and motor recovery (BBS + FMA-LE)

A5: Gait and functional independence (WGS + FIM)

A6: Balance and independence (BBS + FIM)

Statistical Analysis:

Data were processed using SPSS Version 24. Descriptive statistics summarized demographic data. The Kolmogorov-Smirnov test assessed data normality. Paired t-tests and ANOVA were applied to normally distributed data, while Mann-Whitney U and Wilcoxon tests were used for non-parametric comparisons. A p-value < 0.05 was considered statistically significant.

This trial aims to determine which physiotherapy combination is most effective in promoting recovery of walking ability, balance, and independence, with potential implications for developing best-practice rehabilitation protocols for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 80 years
* Both males and females
* Clinically confirmed diagnosis of ischemic or hemorrhagic stroke, verified through CT or MRI (Teodoro et al., 2024)
* At least three months post-stroke to ensure clinical stability
* Residing in the community (not in acute or long-term care facilities)
* Able to understand and follow instructions, assessed by a Glasgow Coma
* Scale (GCS) score of 9 or above (Kim et al., 2021)
* Able to perform basic mobility tasks independently, such as standing, walking short distances, and transferring

Exclusion Criteria:

* Diagnosis of other neurological disorders such as Parkinson's disease or multiple sclerosis
* History of more than one previous stroke
* GCS score below 9, indicating significant cognitive impairment
* Inability to perform basic mobility tasks without assistance
* Presence of severe comorbidities that may impact recovery, such as uncontrolled diabetes or cardiovascular disease
* History of major surgery within the last three months
* Participants in acute or long-term care settings rather than home or community settings (Stephenson et al., 2014; Kim et al., 2022)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Wisconsin Gait Scale (WGS) Scores | Baseline, 3 weeks, and 6 weeks post-intervention
  The WGS evaluates gait deviations in stroke survivors. This outcome assesses improvements in gait pattern, weight transfer, and limb advancement. A lower score post-intervention indicates improved gait function.
Change in Mobility Level (MBL) from the Functional Independence Measure (FIM) | Baseline, 3 weeks, and 6 weeks post-intervention
  The mobility subscale of the FIM assesses transfers, locomotion, and walking independence. A higher score post-treatment indicates reduced caregiver dependence and greater functional mobility.
Change in Lower Extremity Motor Function (LEMF) from the Fugl-Meyer Assessment (FMA-LE) | Baseline, 3 weeks, and 6 weeks post-intervention
  The FMA-LE evaluates reflexes, voluntary movement, coordination, and speed in the lower limbs post-stroke. Improvement in scores reflects enhanced neuromuscular recovery and motor control.

SECONDARY OUTCOMES:
Change in Balance Performance from the Berg Balance Scale (BBS) | Baseline, 3 weeks, and 6 weeks post-intervention
  The BBS assesses static and dynamic balance through 14 tasks such as standing, reaching, and turning. Improved scores indicate better postural control and reduced fall risk in stroke survivors.

OTHER OUTCOMES:
Composite Score Analysis of Combined Functional Measures (A1-A6) | Baseline, 3 weeks, and 6 weeks post-intervention
  To provide a comprehensive evaluation of intervention outcomes, composite scoring analyses will be conducted using six pre-specified combinations of validated tools:
  A1: WGS + FMA-LE + FIM + BBS A2: WGS + BBS A3: WGS + FMA-LE A4: BBS + FMA-LE A5: WGS + FIM A6: BBS + FIM These combinations allow for domain-specific evaluation of gait, motor function, balance, and independence, and will be used to detect multi-domain changes across intervention groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Sehat Medical Complex, Hanjarwal, UOL, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teodoro J, Fernandes S, Castro C, Fernandes JB. Current Trends in Gait Rehabilitation for Stroke Survivors: A Scoping Review of Randomized Controlled Trials. J Clin Med. 2024 Feb 27;13(5):1358. doi: 10.3390/jcm13051358. PMID 38592172
- [Background] Mohan DM, Khandoker AH, Wasti SA, Ismail Ibrahim Ismail Alali S, Jelinek HF, Khalaf K. Assessment Methods of Post-stroke Gait: A Scoping Review of Technology-Driven Approaches to Gait Characterization and Analysis. Front Neurol. 2021 Jun 8;12:650024. doi: 10.3389/fneur.2021.650024. eCollection 2021. PMID 34168608
- [Background] Kim CH, Chu H, Kang GH, Kim KH, Lee YU, Lim HS, Sung KK, Lee S. Comparison of gait recovery patterns according to the paralyzed side in stroke patients: An observational study based on a retrospective chart review (STROBE compliant). Medicine (Baltimore). 2021 Apr 23;100(16):e25212. doi: 10.1097/MD.0000000000025212. PMID 33879656